CLINICAL TRIAL: NCT02877498
Title: A Study to Compare Adaptive Support Ventilation vs. Volume Controlled Ventilation for Management of Respiratory Failure in Patients With Neuroparalytic Snake Envenomation
Acronym: ASV vs VCV in
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Inderpaul singh, Assistant Professor, Department of Pulmonary Medicine, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NK/2194/Study/1241(168)
Record Dates: First submitted 2016-08-17; First posted 2016-08-24 (Estimated); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Snake Envenomation; Invasive Mechanical Ventilation; Adaptive Support Ventilation
MeSH Terms: conditions — Snake Bites

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adaptive support ventilation (Experimental): adaptive support ventilation mode during invasive mechanical ventilation
  Interventions: Other: Adaptive support ventilation
- Volume controlled ventilation (Active Comparator): Volume controlled ventilation during invasive mechanical ventilation
  Interventions: Other: Volume controlled ventilation

INTERVENTIONS:
Other: Adaptive support ventilation — Adaptive support ventilation during invasive mechanical ventilation
  Arms: Adaptive support ventilation
Other: Volume controlled ventilation — Volume controlled ventilation during invasive mechanical ventilation
  Arms: Volume controlled ventilation

SUMMARY:
Neuroparalytic snake envenomation results in severe muscle weakness and respiratory failure. Treatment requires administration of anti-snake venom and supportive care in the form of invasive mechanical ventilation. Whether using adaptive support ventilation (a closed loop mode of ventilation) in comparison to volume controlled ventilation will shorten the duration of ventilation remains undetermined. The current study is planned to compare adaptive support ventilation (ASV) mode of ventilation versus volume controlled ventilation (VCV) during invasive mechanical ventilation for the management of respiratory failure secondary to neuroparalytic snake envenomation.

DETAILED DESCRIPTION:
Snake envenoming is a common medical emergency encountered in the tropical countries, and an estimated 35,000 -50,000 people die of snakebite every year in India. The bites of elapid snakes cause predominantly neurotoxicity, which manifests as ocular and bulbar paralysis, and paralysis of the muscles of respiration, with resultant respiratory failure. The management of these patients includes ventilatory support and administration of snake anti-venom. Respiratory failure requiring mechanical ventilatory support is a frequent cause of admission to the intensive care unit (ICU). Mechanical ventilation is a life-saving intervention, and once there is improvement of the underlying indication, it can be withdrawn abruptly in the majority. However, approximately 20-30% of patients still require gradual discontinuation (ie, weaning). This process is not only difficult in patients with chronic respiratory diseases and acute neuromuscular disorders, such as neurotoxic snake bite, but is also associated with important complications, such as nosocomial pneumonia, prolonged ICU stay, and even mortality, especially in those with persistent weaning failure.

Adaptive support ventilation (ASV) is a closed-loop ventilation mode designed to provide a user-set minimum minute ventilation in intubated patients, either actively breathing or passively ventilated. ASV automatically selects a target ventilatory pattern based on user inputs [patient's predicted body weight (PBW), minimum minute volume, and pressure limit] and respiratory mechanics data from the ventilator monitoring system (respiratory system expiratory time constant and dynamic compliance). The algorithm selects ventilatory parameters so as to minimize total work of inspiration, and the ventilator continuously adapts to match changes in respiratory mechanics by using automatic controls for level of inspiratory pressure above positive end-expiratory pressure (PEEP), frequency, and inspiratory time of ventilator-initiated breaths.

In most studies, ASV has been used only in the weaning phase, and patients were ventilated with conventional modes until weaning. However recent studies suggest its role in primary ventilation in the initial phase of respiratory failure. Previous use of ASV in patients with acute respiratory distress syndrome has been described from our center and the use of ASV was equally efficacious to conventional mode of ventilation (volume control). In another study the use of ASV in comparison to pressure control ventilation in patients with acute respiratory failure reduced the weaning duration and total duration of mechanical ventilation. Because ASV can be used from intubation to extubation, it may also offer some advantages before the weaning phase in patients with respiratory failure. Therefore, we hypothesize that ASV may shorten the total mechanical ventilation (MV) duration, weaning duration, and increase the weaning success rates when compared with conventional ventilation in the management of patients with neuroparalytic snake envenomation.

ELIGIBILITY:
Inclusion Criteria:

1. Need for invasive mechanical ventilation for management of respiratory failure
2. age group of 12 to 90 years
3. ability to provide informed consent to participate in the study

Exclusion Criteria:

1. Cardiorespiratory arrest requiring cardiopulmonary resuscitation
2. pregnancy
3. failure to provide informed consent

Ages: 12 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Liberation from mechanical ventilation | 28 days after discharge
  Liberation from mechanical ventilation (defined as time [in hours] between intubation to extubation for at least six hours)

SECONDARY OUTCOMES:
Incidence of ventilator associated pneumonia | 28 days after discharge
  Ventilator associated pneumonia
Post extubation respiratory failure | 28 days after discharge
  Post extubation respiratory failure (defined as need for either NIV or reintubation)
In hospital mortality | 28 days after discharge
  Death during hospital stay
ICU and hospital length of stay | 28 days after discharge
  Intensive care unit and hospital length of stay

CONTACTS AND LOCATIONS:
Overall Officials: Ritesh Agarwal, MD,DM, Study Director — PGIMER,Chandigarh
Locations (1):
- Respiratory ICU, Post Graduate Institue of Medical Education and Research, Chandigarh, India